CLINICAL TRIAL: NCT05166408
Title: A Novel Technique Predicting Velopharyngeal Insufficiency Risk in Newborns Following Primary Cleft Repair. A Randomised Clinical Trial Comparing Buccinator Flap and Bardach; Two-flap Palatoplasty.
Brief Title: Fistiulation Rate Following Primary Cleft Repair≤
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Walaa Kadry, Lecturer of oral and Maxillofacial Surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Primary palatoplasty fistula
Record Dates: First submitted 2021-12-05; First posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Cleft Palate
Keywords: Cleft palate; Primary repair; Buccinator flap; Palatal fistula
MeSH Terms: conditions — Cleft Palate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buccinator myomucosal flap for primary cleft repair (Other): Study group
  Interventions: Procedure: Buccinator myomucosal flap
- Bardach two flap palatoplasty for primary cleft repair (Other): Control group
  Interventions: Procedure: Bardach two flap palatoplasty

INTERVENTIONS:
Procedure: Buccinator myomucosal flap — Buccinator myomucosal flap for primary cleft palate palatoplasty
  Arms: Buccinator myomucosal flap for primary cleft repair
Procedure: Bardach two flap palatoplasty — Bardach two flap palatoplasty
  Arms: Bardach two flap palatoplasty for primary cleft repair

SUMMARY:
Aim : The aim of present study was to evaluate the buccinator flap utilization in primary cleft palatoplasty on fistulation rate.

Methodology: forty six patients suffering from complete wide cleft palate were randomly divided into two equal groups: study group: the cleft palate defect was repaired by buccinator myomucosal flap whereas the control group patients' clefts were repaired by Bardach (two flap) palatoplasty during primary repair. All patients evaluated at 1 week,3,6 months interval to detect fistulation and measure palatal length by taking impressions and pouring casts to measure palatal length.

DETAILED DESCRIPTION:
Aim : The aim of present study was to evaluate the buccinator flap utilization in primary cleft palatoplasty on fistulation rate. The goal was to predict the risk of velopharyngeal insufficiency and to decrease the fistiulation rate.

Methodology: forty six patients suffering from complete wide cleft palate were randomly divided into two equal groups: study group: the cleft palate defect was repaired by buccinator myomucosal flap whereas the control group patients' clefts were repaired by Bardach (two flap) palatoplasty during primary repair. All patients evaluated at 1 week,3,6 months interval to detect fistulation and measure palatal length by taking impressions and pouring casts to measure palatal length from anterior reference point(incisive foramen) to posterior reference point(uvula) and calculation of change in palatal length.

ELIGIBILITY:
Inclusion Criteria:

1. patients suffering from complete wide cleft palate more than 10 mm
2. Patients age from 9 to 18 months
3. Patients free from any systemic disease that might affect normal healing or the predictable outcome
4. Patients who will agree to the consent and stick to the follow up period

Exclusion Criteria:

1. Patients with systemic disease
2. Patients who might not stick to the follow up period
3. Patients with Pierre Robin syndrome
4. Patients with previous palatal repair

Ages: 9 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Fistiulation rate | 6 months
  The rate of palatal fistula formation following primary cleft palate repair ( number of patients complicated with palatal fistula compared to the full patients number)

SECONDARY OUTCOMES:
Palatal length & risk of VPI | 6 months
  The length of soft palate after surgical repair in correlation with the risk of future velopharyngeal insufficiency ( linear scale)

CONTACTS AND LOCATIONS:
Overall Officials: Wael Abdelsamee, Study Chair — Research organizer
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt